CLINICAL TRIAL: NCT03793816
Title: Tonsillectomy Using BiZact™ - a Randomized Side-controlled Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Assoc. Prof. PD Dr. Gregor Heiduschka, Assoc. Prof. PD M.D., Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EK Nr: 1399/2018
Record Dates: First submitted 2019-01-01; First posted 2019-01-04 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2021-01

CONDITIONS: Tonsillitis Chronic; Tonsillectomy; Hemorrhage; Postoperative Pain; Postoperative Hemorrhage; Surgery--Complications; Handling; Otorhinolaryngologic Diseases
MeSH Terms: conditions — Hemorrhage; Pain, Postoperative; Postoperative Hemorrhage; Otorhinolaryngologic Diseases

STUDY DESIGN:
Intervention Model Description: Cross-over block design with block sizes of 12, such that after 12 patients every group was chosen three times. 48 patients in 4 groups (BiZactTM first / BiZactTM second, BiZactTM right / BiZactTM left side).
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients will not be informed which side was operated with the BiZact™ device. Surgeons however inevitably know side. The side will also be documented in the surgical report. Follow-up specialists must refrain from reading through surgical reports, thus not know which technique was used for which side. Discharging letters will not include technique information.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BiZact™ device (Active Comparator): BiZact™ device will be used appropriately to its purpose to remove one tonsil by:
  * Incision of the anterior palatal arch
  * Locating of the cranial pole of the tonsil
  * Dissection of the tonsil capsule
  * Localized coagulation of bleeding vessels
  * Detaching of the inferior pole from the pharynx tissue
  Interventions: Device: BiZactTM Open Sealer/Divider
- Cold steel dissection (CD) (Active Comparator): Cold steel dissection (CD) with localized cauterization for hemostasis serves as the comparative procedure within each patient (cross-over).
  Interventions: Device: BiZactTM Open Sealer/Divider

INTERVENTIONS:
Device: BiZactTM Open Sealer/Divider — The BiZactTM Open Sealer/Divider creates a seal by application of radiofrequency (RF) electrosurgical energy to blood and lymphatic vessels or tissue bundles interposed between the jaws of the instrument. A cutting blade within the instrument is surgeon-activated to divide tissue. It is a single-use device and will not be reused in other patients.

SUMMARY:
Tonsillectomies are frequently followed by severe postoperative pain, hence high analgetics consumption and prolonged hospitalization. Also, postoperative hemorrhages can be hazardous. Constant evaluation of surgical techniques is paramount to improve safety and cost-effectiveness. Frequently tonsillectomies are performed in cold steel technique. Aim of this study will be the evaluation of handling, surgical time, postoperative pain and postoperative hemorrhage rates using the BiZactTM-Device in comparison to traditional techniques on the contralateral side. In one patient, two different techniques will be used.

The primary objective will be the surgical time. Regardless of surgeon handedness, surgeons will randomly be assigned to either start with the left or right tonsil, and randomly either to start with the BiZact™ Device or with "cold steel" methods.

Additionally, time to stop bleeding, intraoperative blood loss, tonsil mobility, device handling, as well as wound healing will be assessed.

DETAILED DESCRIPTION:
Although stricter indication criteria have been implanted (especially in Austria since 2008), tonsillectomies are still performed very frequently. Post-surgical bleeding can potentially be life-threatening, and occur within 3 weeks after tonsillectomy. A broad survey in Great Britain revealed a postoperative hemorrhage rate in 33.921 patients between 1.5 and 5.4 %, varying on hospital size. Small collectives also showed rates up to 21.7%.

Worldwide, different techniques are used. Generally, "cold" steel and "hot" techniques can be distinguished, although often current-carrying ("hot") and "cold" instruments are used alternately. Postoperative pain seems to be uninfluenced by technique, whereas postoperative hemorrhage rates seem to be higher in "hot" techniques.

LigaSure® is a bipolar "current-carrying" device, which is able to seal vessels. Simultaneously tissue impedance is measured to control energy application. In this way only the required energy levels are applied. Therefore LigaSure® can also be referred as a "softened hot" technique.

In 2005 Lachanas et al. compared the LigaSure®-technique with the "cold" steel technique in 200 patients and found significantly less postoperative pain in favor of the LigaSure®-technique. Postoperative hemorrhage rates were not higher with LigaSure®. Based on the LigaSure®-scissors, Medtronic introduced a device specifically developed and licensed for tonsillectomies (BiZactTM).

Aim of this study will be the evaluation of handling, surgical time, postoperative pain and postoperative hemorrhage rates in comparison to traditional techniques on the contralateral side. In one patient, two different techniques will be used. This side-controlled evaluation of surgical techniques in tonsillectomies has been proven successfully in previous studies.

ELIGIBILITY:
Inclusion Criteria:

* Age 14 and older
* Written informed consent (in case of underage participant also parental informed consent)
* Assigned for Tonsillectomy on both sides due to chronic tonsillitis

Exclusion Criteria:

* History of abscesses in tonsillar region
* Coagulation disorder (as assessed by a coagulation questionnaire and blood results)
* Suspicion of untreated malignancy of any kind
* Planned removal of only one tonsil

Ages: 14 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-10-23 (Actual); Study Completion 2020-12-21 (Actual)

PRIMARY OUTCOMES:
surgical time | 1 hour (intraoperative)
  For the aim of the study surgical time is defined as time from superior mucosal incision to the moment when the removed tonsil is placed on instrument table (recorded by theatre staff - stopwatch).

SECONDARY OUTCOMES:
Time to stop bleeding | 1 hour (intraoperative)
  Time to stop bleeding per side after tonsil removal (recorded by theatre staff - stopwatch)
intraoperative blood loss | 1 hour (intraoperative)
  intraoperative blood loss as measured by A) secretion/blood volume in suction device side separately B) number of used swabs C) swab weight (documented by surgical assistant, side separately at the earliest time point after removal out of the oral cavity - weighing scale provided only for this investigation)
Postoperative pain assessment | Day of surgery until 2 months after surgery
  Postoperative pain assessment A) using a side specific questionnaire (visual analogue scales (VAS-Scale) 0-100mm: differences of more than 16mm can be judged as significant in style of Bijur et al. 2001) on days 0, 1, 3, 5, 7 and 10.
  B) follow-up phone call 2 months after surgery (or in-visit as preferred by the patient) assesses for swallowing difficulties and residual pain in side comparison.
Wound healing | approx. 10 days after surgery
  Wound healing on a VAS-Scales for each side (from 0 very nice tissue / no inflammation to 100mm scale very thick fibrin / strong inflammation as seen by redness/secretion) (evaluated by ENT specialist not familiar with previous randomized side in course of postoperative follow-up visit including review of histological findings)
Tonsil mobility intraoperatively | intraoperative
  Tonsil mobility intraoperatively on a VAS-Scales for each side (from 0 not mobile to 100mm very easy to move)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No
individual participant data (IPD) is not to be shared with third party members

REFERENCES:
- [Background] Österreichische Gesellschaften für Hals-Nasen-Ohren-Heilkunde, Kopf- und Halschirurgie und Kinder- und Jugendheilkunde. Joint recommendation on tonsillectomy. Monatsschrift Kinderheilkunde. 2008;156(3):268-271.
- [Background] Lowe D, van der Meulen J. National Prospective Tonsillectomy Audit. Bulletin of The Royal College of Surgeons of England. 2003;85(10):352-353.
- [Background] Sarny S, Habermann W, Ossimitz G, Schmid C, Stammberger H. Tonsilar haemorrhage and re-admission: a questionnaire based study. Eur Arch Otorhinolaryngol. 2011 Dec;268(12):1803-7. doi: 10.1007/s00405-011-1541-y. Epub 2011 Mar 4. PMID 21373896
- [Background] Dadgarnia MH, Aghaei MA, Atighechi S, Behniafard N, Vahidi MR, Meybodian M, Zand V, Vajihinejad M, Ansari A. The comparison of bleeding and pain after tonsillectomy in bipolar electrocautery vs cold dissection. Int J Pediatr Otorhinolaryngol. 2016 Oct;89:38-41. doi: 10.1016/j.ijporl.2016.07.022. Epub 2016 Jul 26. PMID 27619026
- [Background] Riegler M, Cosentini E. Aktueller Stand der LigaSure®/Atlas®-Technologie zur Gefäßversiegelung in der Allgemeinchirurgie. European Surgery. 2004;36(2):85-88.
- [Background] Lachanas VA, Prokopakis EP, Bourolias CA, Karatzanis AD, Malandrakis SG, Helidonis ES, Velegrakis GA. Ligasure versus cold knife tonsillectomy. Laryngoscope. 2005 Sep;115(9):1591-4. doi: 10.1097/01.mlg.0000172044.57285.b6. PMID 16148700
- [Background] Izny Hafiz Z, Rosdan S, Mohd Khairi MD. Coblation tonsillectomy versus dissection tonsillectomy: a comparison of intraoperative time, intraoperative blood loss and post-operative pain. Med J Malaysia. 2014 Apr;69(2):74-8. PMID 25241816
- [Background] Chettri ST, Bhandary S, Nepal A, et al. A single blind controlled study comparing bipolar elecrocautery tonsillectomy to cold dissection method in pediatric age groups. Health Renaissance. 2014;11(3):270-272.
- [Background] Bijur PE, Silver W, Gallagher EJ. Reliability of the visual analog scale for measurement of acute pain. Acad Emerg Med. 2001 Dec;8(12):1153-7. doi: 10.1111/j.1553-2712.2001.tb01132.x. PMID 11733293
- [Derived] Besser G, Grasl S, Meyer EL, Schnoell J, Bartosik TJ, Brkic FF, Heiduschka G. A novel electrosurgical divider: performance in a self-controlled tonsillectomy study. Eur Arch Otorhinolaryngol. 2022 Apr;279(4):2109-2115. doi: 10.1007/s00405-021-07008-9. Epub 2021 Aug 2. PMID 34338876